CLINICAL TRIAL: NCT02997449
Title: Complete Endosonographic Intrathoracic Nodal Staging of Lung Cancer Patients in Whom Stereotactic Ablative Radiotherapy (SABR), is Considered
Brief Title: Complete Endosonographic Intrathoracic Nodal Staging of Lung Cancer Patients in Whom SABR is Considered
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof J.T. Annema, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: STAGE; 2013_196 (Other: Medical Ethics Review Committee Academic Medical Center)
Record Dates: First submitted 2014-10-17; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Non Small Cell Lung Cancer (NSCLC); Intrathoracic Nodal Staging
Keywords: Non-Small Cell Lung Cancer (NSCLC); Stereotactic ablative radiotherapy (SABR); Intrathoracic nodal staging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC, SABR, nodal staging: Patients with a clinical or pathological diagnosis of Non-Small Cell Lung Cancer (NSCLC), and who are medically inoperable or refuse surgery, are eligible if Stereotactic ablative radiotherapy (SABR) is recommended by a multi-disciplinary tumor board. All patients undergo complete mediastinal and hilar staging procedure (EBUS+EUS-B). Pre endoscopy imaging data will be compared with endosonography data.

SUMMARY:
Rationale: Accurate staging of lung cancer is important because it directs treatment and determines prognosis. The development of Stereotactic Ablative Radiotherapy (SABR), has revolutionized radiation therapy for early stage lung cancer and results demonstrate similar outcomes in comparison to surgical resection of the lung tumor. The staging work-up program for patients with a potentially resectable Non-Small-Cell Lung Cancer (NSCLC) includes at least a computed tomography (CT) scan of the chest and integrated Positron Emission Tomography - Computed Tomography (PET/CT) scans, and when indicated, invasive mediastinal staging. However, patients who are treated with SABR do not routinely undergo the same nodal staging work-up as do surgical candidates. As both surgery and SABR appear to achieve comparable rates of local and regional tumor control, it appears only logical to perform a similar staging work-up in all patients with early stage lung cancer who will be treated with either of the two curative local modalities. In the past, a lack of invasive nodal sampling before SABR was considered acceptable as invasive surgical staging (mediastinoscopy) was widely considered the preferred procedure. However, with minimally invasive and safe endosonography procedures now available, improved pre-treatment staging has become possible for patient groups who are eligible for SABR, including those with significant comorbidities.

Hypothesis: Complete endosonographic (combined endobronchial and esophageal) staging of hilar and mediastinal lymph nodes in patients with (suspected) non-small cell lung cancer (NSCLC) will result in change of loco-regional nodal status in 20% of patients, in comparison to staging by PET-CT alone.

Study population: Patients with either established or suspected early-stage NSCLC who are medically inoperable, or who refuse surgery but are potential candidates for SABR with curative intent (provided no intrathoracic metastases are present). Patients will undergo a single scope complete mediastinal and hilar staging procedure (combined EndoBronchial UltraSound (EBUS) and Transesophageal Endoscopic Ultrasound with EBUS scope (EUS-B)).

ELIGIBILITY:
Inclusion Criteria:

* Proven, or highly suspected, non-small cell lung cancer (NSCLC)
* Absence of distant metastases based on PET-CT
* Stereotactic ablative radiotherapy (SABR) with curative intent is contemplated
* One of the following features based on PET-CT:
* Centrally located clinical T1-T2 N0 tumor
* Peripheral located clinical T2 N0 tumor
* Suspicion of N1- N2 disease based on either size (short axis > 10mm CT) or FDG uptake
* Non-FDG avid primary lung tumor and lymph nodes

Exclusion Criteria:

* Medically operable patients with a resectable lung tumor (unless SABR is the explicit preference of the patients or treating physicians preference).
* Bulky nodal disease based on PET-CT
* Contra-indications for endosonography and / or bronchoscopy
* Pregnancy
* Age under 18
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either established or suspected early-stage NSCLC who are medically inoperable, or who refuse surgery but are potential candidates for stereotactic ablative radiotherapy (SABR) with curative intent (provided no intrathoracic metastases are present)
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with change in nodal status based on imaging compared to nodal status based on endosonography. | 0-6 months
  Prior to endoscopy the nodal status (single outcome measure either N0,N1,N2,N3) will be defined based on (PET) CT imaging. After complete endosonographic staging (EBUS+EUS-B) of the hilus and mediastinum again the nodal status will be defined (single outcome measure either N0,N1,N2,N3) based on endosonography findings.
  The sensitivities, negative predictive values (NPV) and positive predictive values (PPV) for endosonography and PET-CT imaging will be calculated.

SECONDARY OUTCOMES:
Radiotherapy plan based on imaging (prior to endosonography) compared to the radiotherapy plan based on endosonography outcomes. | 1 month
  The radiotherapist will make a radiation plan (Gross Tumor Volume (GTV) primary tumor, internal target volume (ITV) primary tumor and planning target volume (PTV) primary tumor) based on (PET) CT imaging prior to endosonography. After endosonography the radiotherapist will make another radiotherapy plan based on endosonography staging results. The proportions of changed radiotherapy plans per patient basis will be calculated.
Incremental pathological confirmation of the diagnosis of lung cancer in patients with only a clinical diagnosis, following endosonographic staging. | 1 month
Complication rate of a complete endosonographic procedure in this patients group | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Netherlands (3):
  - NKI-AvL, Amsterdam
  - VUMC, Amsterdam
  - UMCN, Nijmegen
- Independent Endoscopy Unit, John Paul II Specialist Hospital, Krakow, Poland